CLINICAL TRIAL: NCT00713973
Title: Comparative Study Between American and Brazilian Protocols for Deep Venous Thrombosis Prophylaxis: a New Proposal
Brief Title: Comparative Study Between Thrombosis Prophylaxis Protocols
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Jorge Lorenzoni Moulim, UNESP
Other Study IDs: upeclin/HC/FMB-Unesp-09
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-07

CONDITIONS: Prophylaxis of Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Submitted to the American protocol for prophylaxis of deep vein thrombosis
- 2: Submitted to the Brazilian protocol for prophylaxis of deep vein thrombosis
- 3: Submitted to the SBCP modified protocol for prophylaxis of deep vein thrombosis

SUMMARY:
Background: Compare the American and Brazilian protocols for prophylaxis of deep vein thrombosis (DVT), seeking to draft a new protocol, more comprehensive and applicable. Methods: A prospective study was conducted over a year, covering 212 patients, comparing the protocols on the stratification of risk of DVT, and the type of prophylaxis indicated. A new protocol was proposed, applied and compared to previous.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent plastic surgery in the Hospital of the Medical School of Botucatu, in the period of one year

Exclusion Criteria:

refusal to participate in the research protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent plastic surgery in the Hospital of the Medical School of Botucatu, in the period of one year.
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2007-06; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JORGE L MOULIM, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- University Hospital of UNESP, Botucatu, São Paulo, Brazil